CLINICAL TRIAL: NCT00829283
Title: Treatment of Obesity and Binge Eating: Behavioral Weight Loss Versus Stepped Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0610001922; R01DK049587 (NIH)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Obesity; Binge Eating
Keywords: Experimental; Comparator
MeSH Terms: conditions — Obesity; Bulimia | interventions — sibutramine; Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard Care
  Interventions: Behavioral: Behavioral Weight Loss
- 2 (Experimental): Stepped-care
  Interventions: Behavioral: Behavioral Weight Loss; Behavioral: Behavioral Weight Loss + Guided self-help Cognitive-behavioral Therapy; Drug: Placebo; Drug: Sibutramine/Orlistat

INTERVENTIONS:
Behavioral: Behavioral Weight Loss — weekly individual sessions for 6 months
Behavioral: Behavioral Weight Loss + Guided self-help Cognitive-behavioral Therapy — weekly BWL sessions for 4 weeks and 6-8 CBT sessions for 5 months
  Arms: 2
Drug: Placebo — One pill daily
  Arms: 2
Drug: Sibutramine/Orlistat — Sibutramine 15 mg daily or Orlistat 120mg TID
  Arms: 2

SUMMARY:
This controlled study will test the effectiveness of a stepped-care approach to a standard behavioral weight loss treatment for obese patients with Binge Eating Disorder (BED). The major question is whether the stepped-care approach, which begins with behavioral weight loss and then follows a decision tree for additional interventions based on early treatment response is superior to standard behavioral treatment.

DETAILED DESCRIPTION:
The stepped-care arm of this study included an obesity medication intervention. At the start of the study, the active medication was sibutramine and was compared to a placebo control. On 10/8/2010, Abbott Laboratories withdrew their obesity drug sibutramine (Meridia) from the market in light of clinical trial data pointing to an increased risk for stroke and myocardial infarction. In response to this event, the investigators submitted an IRB amendment to change the active obesity medication from sibutramine to Orlistat. The IRB amendment was approved on 11/4/2010. The PI received approval from NIH/NIDDK Program Officer Robert Kuczmarski to enact this change.

ELIGIBILITY:
Inclusion criteria:

* Obese (BMI>=30)

Exclusion criteria:

* Medication regimen that represents medical contraindication to sibutramine
* Serious unstable or uncontrolled medical conditions that represent contraindication to sibutramine
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Grilo CM, White MA, Ivezaj V, Gueorguieva R. Randomized Controlled Trial of Behavioral Weight Loss and Stepped Care for Binge-Eating Disorder: 12-Month Follow-up. Obesity (Silver Spring). 2020 Nov;28(11):2116-2124. doi: 10.1002/oby.22975. Epub 2020 Sep 27. PMID 32985114

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Standard Care
  Behavioral Weight Loss: weekly individual sessions for 6 months
- Stepped-care: Stepped-care
  Behavioral Weight Loss: weekly individual sessions for 6 months
  Behavioral Weight Loss + Guided self-help Cognitive-behavioral Therapy: weekly BWL sessions for 4 weeks and 6-8 CBT sessions for 5 months
  Placebo: One pill daily
  Sibutramine/Orlistat: Sibutramine 15 mg daily or Orlistat 120mg TID
Period: Overall Study
Arm/Group | Standard Care | Stepped-care
Started | 39 | 152
Completed | 32 | 127
Not Completed | 7 | 25
Not completed — Lost to Follow-up | 7 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Stepped-care | Total
Number analyzed (Participants) | 39 | 152 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.2) | 48.0 (9.6) | 48.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 104 | 136
  Male | 7 | 48 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  White | 30 | 120 | 150
  Black | 5 | 23 | 28
  Hispanic | 3 | 5 | 8
  Asian | 1 | 1 | 2
  Other | 0 | 3 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.5 (5.7) | 39.4 (6.0) | 38.9 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Reached Binge Eating Remission
Description: Binge Remission (abstinence from binge eating)
Time Frame: 12 months follow-up
Measure: Number; unit: participants
Arm/Group | Standard Care | Stepped-care
Number analyzed (Participants) | 39 | 152
participants | 16 | 65

2. Secondary Outcome: BMI
Description: The body mass index is a value derived from the mass and height of an individual. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m^2.
Time Frame: 12 months follow-up post-treatment
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Standard Care | Stepped-care
Number analyzed (Participants) | 32 | 127
kg/m^2 | 35.9 (6.6) | 37.1 (6.7)

ADVERSE EVENTS:
Arm/Group | Standard Care | Stepped-care
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/152
Other Adverse Events (participants affected / at risk) | 0/39 | 0/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No